CLINICAL TRIAL: NCT05943002
Title: Patient-reported, Health Economic and Psychosocial Outcomes in Friedreich Ataxia
Acronym: PROFA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: German Center for Neurodegenerative Diseases (DZNE) (Other)
Collaborators: McMaster University (Other); Sorbonne University (Other)
Responsible Party: Sponsor
Other Study IDs: GR026
Record Dates: First submitted 2023-03-16; First posted 2023-07-12 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-01

CONDITIONS: Friedreich Ataxia
Keywords: health-related quality of life; economic evaluation; psychosocial health; mobile-health app; Friedreich's Ataxia; Ambulatory assessment
MeSH Terms: conditions — Friedreich Ataxia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The PROFA study is an international, multi-centric observational and validation study to assess the patient-reported, psychosocial and economic outcomes of patients with Friedreich Ataxia (FA). Eligible patients will be recruited from six study centers in Germany, Austria and France. Patients will complete a baseline assessment via face-to-face interviews at the study centers and multiple momentary follow-up assessments via a mobile-health app at home daily to monthly for six months. Study results will gain essential and in-depth insights into the daily life of patients with FA.

DETAILED DESCRIPTION:
There is a lack of knowledge about the patient-reported, psychosocial, and economic impact of Friedreich's Ataxia (FA). The few previous studies were based on small sample sizes and annual cross-sectional data, limiting the generalizability of the results.

Therefore, the PROFA study aims

1. to assess the acceptability, feasibility, and usability of a mobile-health app for the collection of longitudinal real-time data,
2. to determine healthcare costs from a societal perspective that includes informal care productivity losses, to assess associated factors and to analyze the impact of evidence-based treatment on costs,
3. to validate measures of health-related quality of life (HRQoL), to assess patients' HRQoL and its fluctuation over time and identify associated factors,
4. to develop, validate and evaluate a new measure of hearing and speech disabilities' impact on patients' psychosocial health, and
5. to evaluate interaction effects between HRQoL, psychosocial health and economic outcomes in patients with FA.

Thus, the PROFA study will gain a comprehensive understanding of the individual, societal, and economic burden of FA, identifying determinants of health and social life and efficient use of healthcare resources. This is crucial to improve the treatment, care, and everyday life of FA patients and their families.

This validation and observational study will recruit patients from six study centers (Germany, France, and Austria). The data assessment will be based on (i) a baseline assessment via interviews at the study centers and (ii) a subsequent remote momentary data assessment via a mobile-health app on a daily to monthly basis for six months, covering assessments of ataxia severity, HRQoL, psychosocial health, speech and hearing disabilities, health services utilization, and specific health events. Descriptive and multivariate statistics will be used to describe the impact of FA on the patient-reported HRQoL, psychosocial health and economic outcomes.

ELIGIBILITY:
Inclusion Criteria:

* FA confirmed by molecular genetic testing
* Ataxia severity of ≤30 points according to the Scale of the Assessment and Rating of Ataxia (SARA)
* Access to a smartphone or tablet and able to operate the device
* Older than 12 years

Exclusion Criteria:

* Lack of ability to give consent
* Ataxia severity >30 according to the Scale of the Assessment and Rating of Ataxia (SARA)

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients in this study have a Friedreich Ataxia (FA) disease confirmed by molecular genetic testing with disease severity of ≤30 points according to the Scale of the Assessment and Rating of Ataxia. FA is the most common hereditary ataxia in Europe. The genetic mutation that underlies almost all FA cases is a homozygous guanine-adenine-adenine triplet repeat expansion in the ﬁrst intron of the FXN gene, which encodes the mitochondrial protein frataxin. Clinical onset of FA occurs most often around puberty, but in a few cases, symptoms develop in adulthood. FA is characterized by muscle weakness, imbalance, poor coordination, sensory loss, and speech problems. FA could cause wheelchair dependency and reduced life expectancy.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2024-08-31 (Estimated); Study Completion 2024-10-31 (Estimated)

PRIMARY OUTCOMES:
Usability of the mobile-health app as a remote monitoring momentary data assessment tool | Six months
  Completeness of data
Acceptability of the mobile-health app as a remote monitoring momentary data assessment tool | Month 6
  Acceptability is assessed by a self-developed questionnaire (asking patients to rate the app based on user experience)
Total societal costs | Six months
  Aggregated healthcare costs of utilized healthcare services, informal care and productivity losses
Health-related quality of life | Month 1
  Health-related quality of life assessed by the "Patient Reported Outcome Measures for Ataxia" Short-Form (PROM-ATAX), with a score range between 0 to 40 with higher scores indicating lower health-related quality of life
Health-related quality of life | Month 3
  Health-related quality of life assessed by the "Patient Reported Outcome Measures for Ataxia" Short-Form (PROM-ATAX), with a score range between 0 to 40 with higher scores indicating lower health-related quality of life
Health-related quality of life | Month 5
  Health-related quality of life assessed by the "Patient Reported Outcome Measures for Ataxia" Short-Form (PROM-ATAX), with a score range between 0 to 40 with higher scores indicating lower health-related quality of life
Health-related quality of life | Month 6
  Health-related quality of life assessed by the "Patient Reported Outcome Measures for Ataxia" Short-Form (PROM-ATAX), with a score range between 0 to 40 with higher scores indicating lower health-related quality of life
Psychosocial health due to communication handicaps caused by speech and hearing disabilities | Month 1
  Psychosocial impact of hearing and speech disabilities assessed by the "Scale for the psychosocial impact of hearing and speech disabilities in Friedreich Ataxia" (COM-ATAX) with a score range between 0 to 68 (higher scores indicate more difficulties)
Psychosocial health due to communication handicaps caused by speech and hearing disabilities | Month 2
  Psychosocial impact of hearing and speech disabilities assessed by the "Scale for the psychosocial impact of hearing and speech disabilities in Friedreich Ataxia" (COM-ATAX) with a score range between 0 to 68 (higher scores indicate more difficulties)
Psychosocial health due to communication handicaps caused by speech and hearing disabilities | Month 3
  Psychosocial impact of hearing and speech disabilities assessed by the "Scale for the psychosocial impact of hearing and speech disabilities in Friedreich Ataxia" (COM-ATAX) with a score range between 0 to 68 (higher scores indicate more difficulties)
Psychosocial health due to communication handicaps caused by speech and hearing disabilities | Month 4
  Psychosocial impact of hearing and speech disabilities assessed by the "Scale for the psychosocial impact of hearing and speech disabilities in Friedreich Ataxia" (COM-ATAX) with a score range between 0 to 68 (higher scores indicate more difficulties)
Psychosocial health due to communication handicaps caused by speech and hearing disabilities | Month 5
  Psychosocial impact of hearing and speech disabilities assessed by the "Scale for the psychosocial impact of hearing and speech disabilities in Friedreich Ataxia" (COM-ATAX) with a score range between 0 to 68 (higher scores indicate more difficulties)
Psychosocial health due to communication handicaps caused by speech and hearing disabilities | Month 6
  Psychosocial impact of hearing and speech disabilities assessed by the "Scale for the psychosocial impact of hearing and speech disabilities in Friedreich Ataxia" (COM-ATAX) with a score range between 0 to 68 (higher scores indicate more difficulties)
Fluctuation of health-related quality of life | Day one, two and three in months 1
  Change in health-related quality of life measured by the 5-level EQ-5D version (EQ-5D-5L) with a score range between 0 and 1 (higher values indicate higher health-related quality of life)
Fluctuation of health-related quality of life | Day one, two and three in months 3
  Change in health-related quality of life measured by the 5-level EQ-5D version (EQ-5D-5L) with a score range between 0 and 1 (higher values indicate higher health-related quality of life)
Fluctuation of health-related quality of life | Day one, two and three in months 5
  Change in health-related quality of life measured by the 5-level EQ-5D version (EQ-5D-5L) with a score range between 0 and 1 (higher values indicate higher health-related quality of life)
Fluctuation of health-related quality of life | Day one, two and three in months 6
  Change in health-related quality of life measured by the 5-level EQ-5D version (EQ-5D-5L) with a score range between 0 and 1 (higher values indicate higher health-related quality of life)

CONTACTS AND LOCATIONS:
Overall Officials: Bernhard Michalowsky, PD Dr., Principal Investigator — German Center for Neurodegenerative Diseases (DZNE) Rostock/ Greifswald, Germany
Locations (6):
- Klinik für Neurologie, Medizinische Universität Innsbruck, Innsbruck, Austria
- Paris Brain Institute, Paris, France
- Germany (4):
  - Department of Neurology, RWTH Aachen University, Aachen
  - German Center for Neuro-degenerative Diseases (DZNE), Bonn
  - Friedrich-Baur-Institut an der Neurologischen Klinik und Poliklinik, Münich
  - Neurologische Klinik und Hertie-Institut für Klinische Hirnforschung, Universitätsklinik Tübingen, Tübingen

REFERENCES:
- [Derived] Buchholz M, Weber N, Borel S, Sayah S, Xie F, Schulz JB, Reetz K, Boesch S, Klopstock T, Karin I, Schols L, Grobe-Einsler M, Klockgether T, Davies EH, Schmeder M, Nadke A, Michalowsky B. Patient-reported, health economic and psychosocial outcomes in patients with Friedreich ataxia (PROFA): protocol of an observational study using momentary data assessments via mobile health app. BMJ Open. 2023 Aug 1;13(8):e075736. doi: 10.1136/bmjopen-2023-075736. PMID 37527887
- See also: PROFAs project overview description from the German sponsor — https://www.gesundheitsforschung-bmbf.de/de/profa-patientenbezogene-gesundheitsokonomische-und-psychosoziale-outcomes-bei-patientinnen-15284.php
- See also: PROFAs project overview description from the EJPRD — https://www.ejprarediseases.org/profa-patient-reported-health-economic-and-psychosocial-outcomes-in-friedreich-ataxia/